CLINICAL TRIAL: NCT03503253
Title: Transcatheter Leak Closure With Detachable Coils Following Incomplete Left Atrial Appendage Closure Procedures
Acronym: TREASURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCAI_Leak closure
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Left Atrial Appendage Incomplete Closure

STUDY DESIGN:
Intervention Model Description: Prospective, single arm study with consecutive, eligible subject enrollment. All subjects will undergo percutaneous LAA leak closure procedure with detachable coils.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-arm (Other): LAA leak closure using detachable coils; Interlock-35 Fibered IDC Occlusion System, Concerto Helix Detachable Coil System
  Interventions: Device: Interlock-35 Fibered IDC Occlusion System; Device: Concerto Helix Detachable Coil System; Device: Azur Peripheral Coil System

INTERVENTIONS:
Device: Interlock-35 Fibered IDC Occlusion System — Use of detachable coil for LAA leak closure
Device: Concerto Helix Detachable Coil System — Use of detachable coil for LAA leak closure
Device: Azur Peripheral Coil System — Use of detachable coil for LAA leak closure

SUMMARY:
Although the clinical impact of left atrial appendage (LAA) leaks still requires confirmation, the open pouch with residual flow resulting from incomplete LAA closure may promote blood stagnation and thrombus formation, and increase the risk of thromboembolic events. The main purpose of this trial is to evaluate the safety and efficacy of percutaneous leak closure with detachable vascular coils.

DETAILED DESCRIPTION:
Therapies locally targeting the LAA via occlusion, exclusion, or excision have emerged as an alternative and effective approach for stroke prophylaxis in AF patients, especially those with OAC contra-indications. Despite mounting evidence of their safety and efficacy in comparison with standard oral therapy, device-related thrombus and incomplete LAA closure resulting in residual, significant leak may occur, potentially hindering an effective stroke prevention. To date, detachable coils have found a wide range of applications for transcatheter occlusion/embolization procedures (e.g., cerebral aneurysms, pulmonary, renal and cerebral arteriovenous malformations, patent ductus arteriosus, endoleaks). The main purpose of this trial is to evaluate the feasibility and efficacy of transcatheter leak closure with detachable coils in patients with evidence of incomplete percutaneous/epicardial LAA exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Presence of a significant LAA leak (moderate/severe following percutaneous occlusions or mild/severe after epicardial exclusions with the LARIAT suture delivery device).
* Less moderate embolic risk (CHA2DS2-VASc ≥2)
* High associated hemorrhagic risk (HASBLED ≥ 3), or absolute contraindication to OAC, or need for prolonged dual antiplatelet therapy, or history of thromboembolic events despite LAA occlusion/exclusion after other potential causes.
* written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Life expectancy < 2 years.
* pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 7 days
  Procedural success, defined as successful delivery, deployment release of detachable coil(s) into the LAA, and incidence of LAA occlusion as measured by fluoroscopy and echocardiographic color Doppler jets less than 3mm by TEE at the end of the procedure.
Rate of LAA leak closure | 60 days
  LAA occlusion will be assessed by TEE color Doppler and will be defined as absence of flow in the LAA or minimal color Doppler jets (< 1mm).
Incidence of Major Adverse Events (MAE) | 30 days
  Rate of procedure- and device-related complications (device embolization; cardiac injury, re-intervention, and/or device-related surgery; bleeding events such as pericardial effusion requiring drainage, cranial bleeding due to any source, gastrointestinal bleeding; transient ischemic attack/stroke; systemic embolism; death; or any other event related to the device or the procedure, which requires treatment).

SECONDARY OUTCOMES:
Composite of all-cause mortality, stroke and bleeding | 12 months
  Composite: stroke or transient ischemic attack, systemic embolism, major bleeding event.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- Texas Cardiac Arrhythmia Institute, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan yet

REFERENCES:
- [Derived] Della Rocca DG, Horton RP, Di Biase L, Bassiouny M, Al-Ahmad A, Mohanty S, Gasperetti A, Natale VN, Trivedi C, Gianni C, Burkhardt JD, Gallinghouse GJ, Hranitzky P, Sanchez JE, Natale A. First Experience of Transcatheter Leak Occlusion With Detachable Coils Following Left Atrial Appendage Closure. JACC Cardiovasc Interv. 2020 Feb 10;13(3):306-319. doi: 10.1016/j.jcin.2019.10.022. Epub 2020 Jan 15. PMID 31954677